CLINICAL TRIAL: NCT01561430
Title: Assessment of Safety, Tolerability, and Pharmacodynamic Effects of LY2886721 in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease
Brief Title: Study of LY2886721 in Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to abnormal liver biochemical tests in some participants.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13735; I4O-MC-BACC (Other: Eli Lilly and Company); 2011-005217-37 (EudraCT Number)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Alzheimer's Disease
Keywords: beta-secretase inhibitor
MeSH Terms: conditions — Alzheimer Disease | interventions — N-(3-(2-amino-4a,5,7,7a-tetrahydro-4H-furo(3,4-d)(1,3)thiazin-7a-yl)-4-fluorophenyl)-5-fluoropicolinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 15 mg LY2886721 (Experimental): LY2886721: 15 milligrams (mg), capsules, administered orally, once daily for 26 weeks.
  Interventions: Drug: LY2886721
- 35 mg LY2886721 (Experimental): LY2886721: 35 mg, capsules, administered orally, once daily for 26 weeks.
  Interventions: Drug: LY2886721
- 70 mg LY2886721 (Experimental): LY2886721: 70 mg, capsules, administered orally, once daily for 26 weeks.
  Interventions: Drug: LY2886721
- Placebo (Placebo Comparator): Placebo: 1 placebo capsule, administered orally, once daily for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2886721
  Arms: 15 mg LY2886721; 35 mg LY2886721; 70 mg LY2886721
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this Phase 1/Phase 2 study is to evaluate how the body handles the drug and the drug's effect on the body of participants with mild cognitive impairment (MCI) due to Alzheimer's Disease (AD) or mild AD and who test positive for amyloid plaque.

ELIGIBILITY:
Inclusion Criteria:

Meets criteria for MCI due to AD or Mild AD

All participants will be required to undergo assessment via the Mini Mental State Examination (MMSE) scale at screening

* Participants with MMSE scores of 20 to 26, inclusive, may be enrolled provided they meet the criteria for mild AD, as follows:

  * Participant meets the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable AD
  * Clinical Dementia Rating Scale (CDR) score of 0.5 or 1
  * Positive scan for the presence of amyloid beta
* Participants with MMSE of 27 to 30, inclusive, may be enrolled as participants with MCI due to AD provided they meet the following criteria:

  * Gradual and progressive change in memory function as reported by the participant or a caregiver during a period of more than 6 months
  * Free and Cued Selective Reminding Test with Immediate Recall (FCSRT-IR): free recall ≤22 and total recall ≤46
  * Absence of dementia
  * Preservation of functional independence
  * Exclusion of other potential (vascular, traumatic, or medical) causes of cognitive decline, where possible
  * Positive scan for the presence of amyloid beta
* Women must be postmenopausal
* Men are required to use an approved barrier method of contraception if their partners are pregnant, or of childbearing potential and not using approved contraceptive methods

Exclusion Criteria:

* Participant in another drug or device study
* Have a history of frontotemporal dementia, Lewy body disease, vascular dementia, Huntington's disease, Parkinson's disease, progressive supranuclear palsy (PSNP), or other movement disorder
* Participants are not on a stable standard of care (acetylcholinesterase inhibitors, memantine) initiated less than 2 months prior to entry or have less than 4 weeks of stable therapy. Note: Stable standard of care is allowed.
* Have had a serious infectious disease affecting the brain in the past 5 years
* Have had a serious or repeat head injury
* Have significant retinal impairment or disease
* Have had a stroke or other circulation problems that are affecting current health
* Have had a seizure
* Have major depressive disorder and are not on a stable dose of medication. Participants who no longer meet the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV) criteria for major depression may be included
* History of schizophrenia, bipolar disorder, or severe mental illness
* History of alcohol or drug abuse
* Have asthma, chronic obstructive pulmonary disease (COPD), or other breathing disease that is not controlled with medicine
* Have human immunodeficiency virus (HIV) or syphilis
* Are taking blood thinners

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- United States (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sun City, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Delray Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quincy, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monroe, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Biella
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam, Netherlands
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Getafe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sant Cugal Del Valles

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As a result of findings from the I4O-MC-BACJ study (NCT01534273), enrollment was discontinued to the 15 milligrams (mg) arm. The 9 participants already enrolled were allowed to continue study treatment at the 15 mg dose.
Period: Overall Study
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Started | 9 | 23 | 18 | 20
Received at Least One Dose of Study Drug | 9 | 23 | 18 | 20
Completed | 8 | 8 | 1 | 7
Not Completed | 1 | 15 | 17 | 13
Not completed — Adverse Event | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 1 | 14 | 13 | 12

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo | Total
Number analyzed (Participants) | 9 | 23 | 18 | 20 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.59 (7.569) | 72.50 (8.378) | 70.23 (8.603) | 67.73 (7.126) | 69.66 (8.201)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 7 | 11 | 33
  Male | 4 | 13 | 11 | 9 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 3 | 0 | 6
  Black or African American | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 9 | 20 | 15 | 20 | 64
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 19 | 15 | 18 | 60
  Netherlands | 1 | 1 | 1 | 2 | 5
  Japan | 0 | 3 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Weeks in Cerebrospinal Fluid (CSF) Amyloid Beta (Aβ)1-40 and Aβ1-42 Concentrations
Description: Percent change in lumbar CSF concentrations of Aβ1-40 and Aβ1-42 from baseline at 12 weeks post-dose was calculated. The units for CSF were picograms per milliliter (pg/mL). Least Squares (LS) means of percent change in concentration from baseline was calculated using analysis of covariance (ANCOVA) with baseline as a covariate and treatment as a fixed effect.
Time Frame: Baseline, 12 weeks
Population: All randomized participants with evaluable post-baseline CSF Aβ1-40 or Aβ1-42 data.
Measure: Least Squares Mean (Standard Error); unit: percent change in Aβ1-40 and Aβ1-42
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Number analyzed (Participants) | 7 | 9 | 5 | 12
percent change in Aβ1-40 and Aβ1-42
  Aβ1-40: number analyzed (Participants) | 7 | 9 | 5 | 11
  Aβ1-40 | -31.8 (7.35) | -57.7 (6.67) | -58.9 (8.73) | 3.7 (5.96)
  Aβ1-42 | -34.4 (7.27) | -52.0 (6.80) | -60.7 (8.42) | 6.5 (6.06)

2. Primary Outcome: Change From Baseline to 26 Weeks in CSF Aβ1-40 and Aβ1-42 Concentrations
Description: Percent change in lumbar CSF concentrations of Aβ1-40 and Aβ1-42 from baseline at 26 weeks post-dose was to be calculated. The units for CSF were picograms per milliliter (pg/mL). LS means of percent change in concentration from baseline was calculated using ANCOVA with baseline as a covariate and treatment as a fixed effect.
Time Frame: Baseline, 26 weeks
Population: Zero participants analyzed. CSF Aβ1-40 and Aβ1-42 concentrations data was not collected for analysis at 26 weeks.
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Plasma Amyloid Beta (Aβ)1-40 and Aβ1-42 Concentrations
Description: Percent change in plasma concentrations of Aβ1-40 and Aβ1-42 from baseline at 12 weeks and 26 weeks post-dose was calculated. The units for CSF were picograms per milliliter (pg/mL).
Time Frame: Baseline, 12 weeks, 26 weeks
Population: All randomized participants with evaluable post-baseline CSF Aβ1-40 or Aβ1-42 data.
Measure: Mean (Standard Deviation); unit: percent change in Aβ1-40 and Aβ1-42
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Number analyzed (Participants) | 6 | 8 | 4 | 12
percent change in Aβ1-40 and Aβ1-42
  Aβ1-40, Week 12 | -73.4 (6.22) | -80.8 (8.07) | -88.1 (2.66) | 1.90 (15.0)
  Aβ1-40, Week 26: number analyzed (Participants) | 5 | 6 | 1 | 6
  Aβ1-40, Week 26 | -72.3 (11.5) | -85.0 (3.89) | -89.1 (NA) — Standard deviation not reported due to not enough participants for analyses. | 0.944 (22.6)
  Aβ1-42, Week 12 | -63.4 (6.11) | -71.1 (8.38) | -78.2 (5.08) | 0.541 (10.1)
  Aβ1-42, Week 26: number analyzed (Participants) | 5 | 6 | 1 | 6
  Aβ1-42, Week 26 | -65.1 (8.85) | -75.0 (4.33) | -80.8 (NA) — Standard deviation not reported due to not enough participants for analyses. | 1.82 (9.98)

4. Secondary Outcome: Change From Baseline to 26 Weeks in Neuropsychological Test Battery (NTB)
Description: The NTB is a composite cognitive measure in clinical Alzheimer's disease studies and is a collection of several written and oral tests that examines verbal and nonverbal brain functions. NTB Z-score typically ranges from -3 to 3, with lower scores suggesting greater cognitive impairment. LS means were calculated using ANCOVA with baseline as a covariate and treatment as a fixed effect.
Time Frame: Baseline, 26 weeks
Population: All randomized participants with evaluable NTB data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Number analyzed (Participants) | 8 | 7 | 1 | 9
units on a scale | -0.039 (0.1096) | -0.161 (0.1165) | 0.424 (0.3156) | -0.262 (0.1028)

5. Secondary Outcome: Change From Baseline to 26 Weeks in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)
Description: ADAS-Cog11 is an 11-item instrument measuring impairment in memory (Items 1-4, 7, 11), praxis (Items 4 and 5), orientation (Item 6), and language (Items 8-10). Item 1 ranged 0 (all items recalled correctly)-10 (none recalled correctly); Items 2-5 and 8-11 ranged 0 (all items named, performed, drawn, spoken, remember correctly/clearly)-5 (none correct/not clearly spoken); Item 6 ranged 0 (no incorrect responses)-8 (all incorrect); and Item 7 ranged 0 (all words remembered correctly)-12 (no words remembered correctly) for a total ADAS-Cog11 score of 0-70 with higher scores indicating greater disease severity. A score of 0-10 for delayed free recall and a conversion code of 0-5 for digit cancellation and maze completion was added to the total ADAS-Cog11 score for a total ADAS-Cog14 score ranging 0-90 with higher scores indicating greater impairment. LS means were calculated using Mixed Model Repeated Measures (MMRM) with Treatment + Visit + Treatment*Visit + Baseline + Baseline*Visit.
Time Frame: Baseline, 26 weeks
Population: All randomized participants with evaluable ADAS-Cog data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Number analyzed (Participants) | 7 | 9 | 1 | 9
units on a scale | 1.1 (2.77) | 0.6 (2.48) | 0.6 (7.41) | 1.3 (2.44)

6. Secondary Outcome: Change From Baseline to 26 Weeks in the Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB)
Description: The CDR-SB is a composite measure of 6 domains of cognitive and functional performance: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Scores ranged from 0 to 18, with higher scores indicating greater impairment. LS means were calculated using MMRM with Treatment + Visit + Treatment*Visit + Baseline + Baseline*Visit.
Time Frame: Baseline, 26 weeks
Population: All randomized participants with evaluable CDR-SB data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Number analyzed (Participants) | 8 | 9 | 1 | 8
units on a scale | 0.80 (0.432) | 0.52 (0.395) | 1.50 (1.013) | 1.19 (0.402)

7. Secondary Outcome: Change From Baseline to 26 Weeks in Mini Mental State Examination (MMSE)
Description: The MMSE (Folstein et al. 1975) is one of the most widely used screening instruments for cognitive impairment. The test consists of five sections (orientation, registration, attention-calculation, recall, and language) and provides a total score ranging from 0 to 30, with lower scores indicative of greater cognitive impairment. LS means were calculated using MMRM with Treatment + Visit + Treatment*Visit + Baseline + Baseline*Visit.
Time Frame: Baseline, 26 weeks
Population: All randomized participants with evaluable MMSE data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- 70 mg LY2886721: 70 mg, capsules, administered orally, once daily for 26 weeks.
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Number analyzed (Participants) | 8 | 9 | 1 | 10
units on a scale | -0.7 (0.87) | -1.8 (0.81) | 0.2 (2.41) | -3.0 (0.77)

8. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Tau and Phosphorylated Tau (Ptau)-181 Concentrations
Description: Percent change in lumbar CSF tau and ptau-181 concentrations from baseline at 12 weeks post-dose and 26 weeks post-dose was calculated. The units for CSF were picograms per milliliter (pg/mL). Least Squares (LS) means of percent change in concentration from baseline was calculated using analysis of covariance (ANCOVA) with baseline as a covariate and treatment as a fixed effect.
Time Frame: Baseline, 12 weeks, 26 weeks
Population: All randomized participants at 12 weeks with evaluable post-baseline CSF Tau or Ptau data.
  Zero participants analyzed for 26 week CSF Tau or Ptau as data was not collected for analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change in tau and ptau-181
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Number analyzed (Participants) | 7 | 9 | 5 | 12
percent change in tau and ptau-181
  CSF Tau, Week 12 | 14.3 (6.06) | 2.6 (5.42) | 6.8 (7.49) | -4.4 (4.63)
  CSF Tau, Week 26: number analyzed (Participants) | 0 | 0 | 0 | 0
  CSF Ptau, Week 12 | 0.7 (4.81) | 1.7 (4.01) | 4.3 (5.41) | -3.6 (3.40)
  CSF Ptau, Week 26: number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- 15 mg LY2886721: LY2886721: 15 mg, capsules, administered orally, once daily for 26 weeks.
Arm/Group | 15 mg LY2886721 | 35 mg LY2886721 | 70 mg LY2886721 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/23 | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 8/9 | 13/23 | 16/18 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg LY2886721 (N=9) | 35 mg LY2886721 (N=23) | 70 mg LY2886721 (N=18) | Placebo (N=20)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg LY2886721 (N=9) | 35 mg LY2886721 (N=23) | 70 mg LY2886721 (N=18) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colour vision tests abnormal red-green (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram change (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apraxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased vibratory sense (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypnopompic hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obsessive thoughts (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parasomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep talking (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stereotypy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early because of abnormal liver biochemical tests levels for 4 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days